CLINICAL TRIAL: NCT00570258
Title: Randomized, Double Blind Multicenter Phase II Study of Time to Progression on Fulvestrant in Combination With Erlotinib or Placebo in Hormone Receptor-Positive Metastatic Breast Cancer (MBC) Subjects Who Progressed on First Line Hormonal Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA approved higher dose of study drug. Dose used in protocol lower than SOC - enrollment stopped, those on treatment were given option to opt out.
Sponsor: University of Arkansas (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 57485; UARK 2004-19 (Other: UAMS)
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2 (Placebo Comparator): Fulvestrant: 250 mg IM Q 4 weeks
  Placebo: 150 mg PO QD
  Interventions: Drug: Fulvestrant; Drug: Placebo
- 1 (Active Comparator): Fulvestrant: 250 mg IM Q 4 weeks
  Erlotinib: 150 mg PO QD
  Interventions: Drug: Fulvestrant; Drug: erlotinib

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant: 250 mg IM Q 4 weeks
  Arms: 1
Drug: erlotinib — 150 mg PO QD
  Arms: 1
Drug: Fulvestrant — 250 mg IM Q 4 weeks
  Arms: 2
Drug: Placebo — Placebo 150 mg PO QD
  Arms: 2

SUMMARY:
This is a multicenter, randomized, double-blind study of fulvestrant plus erlotinib versus fulvestrant plus placebo for subjects with metastatic breast cancer whose disease progression after first line hormonal therapy.

1. To obtain preliminary estimates of the magnitude and variability of the efficacy of fulvestrant in combination with erlotinib in this subject population, and
2. To obtain historically up-to-date estimates of the magnitude and variability of the efficacy of fulvestrant as the sole active agent in this subject population.

The measure of efficacy for both primary objectives will be time to progression.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind study of fulvestrant plus erlotinib versus fulvestrant plus placebo for subjects with metastatic breast cancer whose disease progressed after first line hormonal therapy.

* Total number of subjects planned for the trial is 130 subjects, that is, approximately 65 subjects in each arm.
* Subjects will be randomized to receive fulvestrant/erlotinib (arm A) or fulvestrant/placebo (arm B) and stratified based on accrual center.
* The study is a parallel-arm double-blind study, with fulvestrant + placebo on the monotherapy arm, and fulvestrant + erlotinib on the combination arm.
* The primary variable outcome is time to progression.
* Subjects whose metastatic disease was diagnosed more than 12 months after completing adjuvant hormonal therapy are eligible to this study if their breast cancer is hormone-receptor-positive and after disease progression on first line hormonal therapy in the metastatic setting. Subjects may have received no more than one line of chemotherapy. While receiving one line of hormonal therapy in the metastatic setting is a requirement, receiving chemotherapy is not, and one line of chemotherapy in the metastatic setting would not exclude these subjects from the trial. Subjects who had a recurrence while on adjuvant hormonal treatment or within 12 months of completion of the adjuvant hormonal treatment are also eligible without the need to receive first line hormonal therapy in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign a written consent.
2. Subjects must have estrogen- and/or progesterone-receptor-positive histologically confirmed adenocarcinoma of the breast with recurrent or metastatic carcinoma of the breast.
3. Baseline measurements and evaluations of involved sites should be performed as close as possible to study entry, but must be within 4 weeks prior to randomization.
4. Subjects fulfilling one of the following criteria are eligible to participate in the study: Subjects with measurable disease as per RECIST criteria. This is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as over 20 mm with conventional technique or as over 10 mm with spiral CT scan or MRI. Subjects with bone lesions, lytic or mixed (lytic + sclerotic), in the absence of measurable disease as defined by RECIST criteria. The lytic component of at least one bone lesion should measure 20 mm with conventional techniques or 10 mm with spiral CT scan or MRI. At least one bone lesion satisfying these criteria must be outside any previously irradiated area.
5. All subjects must be postmenopausal females defined by:

Prior bilateral oophorectomy OR No menstrual period for 12 months or longer. If age 55 years or less and on tamoxifen within the prior 6 months, must have an estradiol level in the postmenopausal range.

Exclusion Criteria:

1. Subjects must not have had more than 1 prior chemotherapy regimen for metastatic disease and no chemotherapy within 3 weeks prior to randomization. 2. No concurrent chemotherapy is allowed while on protocol therapy. Subjects whose adjuvant hormonal therapy was discontinued more than 12 months ago must have had only 1 prior hormonal therapy for metastatic disease. Subjects who relapsed while receiving adjuvant hormonal therapy or less than 12 months after completing adjuvant hormonal therapy may be enrolled directly in the trial.

3. No prior therapy with an estrogen receptor down-regulator (e.g. fulvestrant). Non-protocol concurrent hormonal therapy is not allowed. Subjects must not have had prior therapy with agents that target EGFR. Previous, but not concomitant, therapy with trastuzumab (Herceptin) is allowed. Subjects must not receive trastuzumab (Herceptin) within 3 weeks prior to randomization.

4. Subjects must have ECOG performance status of 0, 1, or 2. 5. Subjects must have adequate hematologic, hepatic, and renal function defined by the following within 4 weeks prior to randomization: Neutrophils > 1500/mm3 and platelets over 100,000/mm3 Total Bilirubin under 1.25 x Institutional upper limit of normal SGPT (ALT) and SGOT (AST) under 2.5 x Institutional upper limit of normal if no demonstrable liver metastases or under 5 x Institutional upper limit of normal in the presence of liver metastases Calculated creatinine clearance over 30ml/min using the following formula: Ccr = (140 - age in years) times (weight in kgs) times 0.085 72 x serum creatinine in mg/dL INR, PT and PTT under 1.5 x Institutional upper limit of normal.

6. Subjects must not be receiving therapy with anticoagulants or have other contraindication to IM injections.

7. Subjects must be age over 18 years. 8. Subjects must not have a history of central nervous system metastasis. 9. Subjects may receive concurrent radiation therapy to painful sites of bony disease or areas of impending fracture as long as the radiation therapy is initiated prior to study entry and sites of measurable disease outside the radiation therapy port are available to follow.

10. Subjects must not take the following medications while enrolled in this trial: ketoconazole, erythromycin, verapamil.

11. Subjects age less than 55 years must not be receiving LHRH agonists or antagonists within 3 months prior to randomization.

12. Subjects who have an ocular inflammation or infection should be fully treated before entry into the trial.

13. Subjects with a neuropathic keratopathy or diabetes or those with anterior basement membrane disease must be advised of the need for frequent ophthalmologic exams.

14. Subjects who continue to wear contact lenses must be advised that they have an increased risk of ocular events. The decision to wear contact lenses should be discussed with the patient's treating oncologist and ophthalmologist.

15. Subjects must not suffer from medical or psychiatric conditions that would interfere with protocol compliance, the ability to provide informed consent, or assessment of response or anticipated toxicities.

16. Subjects must be disease-free of prior invasive malignancies for over 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Makhoul, MD, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - NEA Clinic, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands oncology Group, Springdale, Arkansas
  - Emory University, Atlanta, Georgia
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - Hackensack University, Hackensack, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant Plus Placebo: Fulvestrant: 250 mg IM Q 4 weeks
  Placebo: 150 mg PO QD
  Fulvestrant: 250 mg IM Q 4 weeks
  Placebo: Placebo 150 mg PO QD
- Fulvestrant Plus Erlotinib: Fulvestrant: 250 mg IM Q 4 weeks
  Erlotinib: 150 mg PO QD
  Fulvestrant: Fulvestrant: 250 mg IM Q 4 weeks
  erlotinib: 150 mg PO QD
Period: Overall Study
Arm/Group | Fulvestrant Plus Placebo | Fulvestrant Plus Erlotinib
Started | 12 | 15
Completed | 0 (Early termination due to a change in drug FDA approval.) | 0 (Early termination due to a change in drug FDA approval.)
Not Completed | 12 | 15

BASELINE CHARACTERISTICS:
Population: Early termination due to a change in drug FDA approval. No subject completed study. No data analysis was completed.
Groups:
- Fulvestrant Plus Erlotnib: Fulvestrant: 250 mg IM Q 4 weeks
  Erlotinib: 150 mg PO QD
  Fulvestrant: Fulvestrant: 250 mg IM Q 4 weeks
  erlotinib: 150 mg PO QD
- Total: Total of all reporting groups
Arm/Group | Fulvestrant Plus Placebo | Fulvestrant Plus Erlotnib | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 15 | 21
  >=65 years | 6 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival
Description: This will be defined as the date from randomization onset to first documented occurrence of PD. Death will be regarded as a progression event in those subjects who die before disease progression. Subjects without documented objective progression at the time of the final analysis will be censored at the date of their last tumor assessment.
Time Frame: through study completion, an average of 3 years
Population: Early termination due to a change in drug FDA approval. No subject completed study. No data analysis was completed. No data collected.
Groups:
- Fulvestrant Plus Placebo: Fulvestrant plus placebo: Fulvestrant will be given on day 1 by intramuscular (IM) injection into your buttock muscle(s) then every 28 days. In addition, placebo will be given as a pill, which will be taken by mouth once a day, about the same time of day every day, one hour before or two hours after a meal.
- Fulvestrant Plus Erlotinib: Fulvestrant plus erlotinib: Fulvestrant will be given on day 1 by intramuscular (IM) injection into your buttock muscle(s) then every 28 days. In addition, erlotinib will be given as a pill, which will be taken by mouth once a day, about the same time of day every day, one hour before or two hours after a meal.
Arm/Group | Fulvestrant Plus Placebo | Fulvestrant Plus Erlotinib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants Achieving Either Complete Response or Partial Response
Description: evaluate response rate and the clinical benefit of fulvestrant alone or in combination with erlotinib
Time Frame: through study completion, an average of 3 years
Population: Early termination due to a change in drug FDA approval. Outcome measures not computed on collected data because data would not be statistically relevant. No data analysis was completed. No data collected.
Arm/Group | Fulvestrant Plus Placebo | Fulvestrant Plus Erlotinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Fulvestrant Plus Placebo | Fulvestrant Plus Erlotinib
All-Cause Mortality (participants affected / at risk) | 8/12 | 3/15
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/15
Other Adverse Events (participants affected / at risk) | 3/12 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Plus Placebo (N=12) | Fulvestrant Plus Erlotinib (N=15)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
fever of unknown origin (Immune system disorders) | 0 (0) | 1 (1)
possible heart failure (Cardiac disorders) | 1 (1) | 0 (0)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypotension (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Plus Placebo (N=12) | Fulvestrant Plus Erlotinib (N=15)
anorexia (General disorders) | 1 (1) | 1 (2)
alopecia (General disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6)
fatigue (General disorders) | 1 (1) | 2 (5)
nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 2 (7)
pain (General disorders) | 1 (1) | 5 (5)
dizziness (General disorders) | 1 (1) | 0 (0)
cough (General disorders) | 1 (1) | 0 (0)
bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
pruritis (General disorders) | 0 (0) | 1 (1)
dyspnea (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to a change in drug FDA approval. Outcome measures not computed because data would not be statistically relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No